CLINICAL TRIAL: NCT05812339
Title: Body Surface Gastric Mapping to Evaluate Patients With Upper Gastrointestinal Symptoms and Controls
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1925
Record Dates: First submitted 2023-02-13; First posted 2023-04-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Motility Disorder; Gastroparesis; Functional Dyspepsia; Cyclical Vomiting; Cannabinoid Hyperemesis Syndrome; Diabetic Gastroparesis
MeSH Terms: conditions — Gastroparesis; Familial cyclic vomiting syndrome; Cannabinoid Hyperemesis Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Motility Disorder Patients: Adults with history of confirmed motility disorder.
  Interventions: Device: Gastric Alimetry System
- Healthy Controls: Adults meeting all inclusion and exclusion criteria with no symptoms or history of motility disorder.
  Interventions: Device: Gastric Alimetry System

INTERVENTIONS:
Device: Gastric Alimetry System — Gastric Alimetry is a medical device intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of gastrointestinal motility disorders. The device is indicated for use during the diagnostic work-up of patients reporting gastric symptoms, who are suspected of having an underlying gastric motility problem.

SUMMARY:
This is an analytical validation observational cohort study is designed to provide evidence of: safety and reliability of Body Surface Gastric Mapping using the Gastric Alimetry System (GAS), normal reference values, and correlation of metrics with patient symptoms among healthy adults and patients diagnosed with upper abdominal motility disorders.

GAS is intended to record, store, view and process gastric myoelectrical activity. This is a proprietary system consisting of multiple electrodes arranged on an array that is placed precisely over the stomach, a reader to collect the electrode measurements and a smart tablet application to track patient reported symptoms. Participants meeting inclusion and exclusion criteria will continue fasting for 30 minutes after the Gastric Alimetry System has been applied and begun measuring, eat a standard study meal within 10 minutes and remain quietly seated, reclining, for 4 hours as the GAS continues to collect data. The array is removed and the abdomen is examined for evidence of skin effects.

ELIGIBILITY:
Inclusion Criteria:

Healthy Population:

* Adults aged 18 years and over
* Able to understand the risks/benefits of the study
* Able to give written informed consent
* No active gastrointestinal symptoms or pathology
* Resides in the Calgary, Alberta area

Patient Population:

* Adults aged 18 years and over
* BMI > 35
* Able to understand the risks/benefits of the study
* Able to give written informed consent
* Patients meeting Rome IV Criteria for functional dyspepsia, or a nausea and vomiting disorder
* Patients with gastroparesis defined on a standardized gastric scintigraphy study
* Resides in the Calgary, Alberta area

Exclusion Criteria:

Healthy Population:

* Under 18 years of age
* BMI > 35
* Taking medications known to affect GI motility or the mid-gut axis (eg antidepressants, anti-anxiety medication, prokinetics, opiates)
* Metabolic, neurogenic, or endocrine disorders known to cause gastrointestinal dysmotility (eg. Multiple Sclerosis, Parkinson's disease, hypothyroidism)
* Known current GI infection (includes H. pylori when being actively treated)
* Known current inflammatory bowel disease
* Known current GI malignancy
* Known GI functional or motility disorders
* Previous gastroduodenal surgery
* GI functional or motility disorders
* Pregnant women
* Open abdominal wounds or abdominal skin not intact (eg rash, abrasions, weeping tissue)
* Fragile skin evidence by high susceptibility to skin tears or skin that bruises and breaks easily
* Allergy to adhesives
* History of allergy or intolerance to ingredients in the meal (nutrient drink, Ensure or similar and Clif bar or similar)
* No vulnerable groups such as; prisoners, individuals with known cognitive impairment, or institutionalised individuals be involved
* Regular cannabis use
* Diagnosed with, or suspected to have life-threatening conditions that could result in immediate danger

Patient Population:

* Under 18 years of age
* BMI > 35
* Metabolic, neurogenic, or endocrine disorders known to cause gastrointestinal dysmotility (eg. Multiple Sclerosis, Parkinson's disease, hypothyroidism)
* Known current GI infection (includes H. pylori when being actively treated)
* Known current inflammatory bowel disease
* Known current GI malignancy
* Previous gastroduodenal surgery
* Open abdominal wounds or abdominal skin not intact (eg rash, abrasions, weeping tissue)
* Fragile skin evidence by high susceptibility to skin tears or skin that bruises and breaks easily
* Allergy to adhesives
* Pregnant women
* History of allergy or intolerance to ingredients in the meal (nutrient drink, Ensure or similar and Clif bar or similar)
* No vulnerable groups such as; prisoners, individuals with known cognitive impairment, or institutionalised individuals be involved
* Regular cannabis use except in the case of CHS
* Diagnosed with, or suspected to have life-threatening conditions that could result in immediate danger
* Inability to remain in a relaxed reclined position for the test duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in the Calgary Alberta region.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric electrical signal frequency | Pre-meal
  Successful detection of gastric electrical signal in the 2-5 cycle-per-minute (cpm) spectrum as defined by reference ranges at Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal frequency | Post meal at 1 hour
  Successful detection of gastric electrical signal in the 2-5 cycle-per-minute (cpm) spectrum as defined by reference ranges at Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal frequency | Post meal at 2 hours
  Successful detection of gastric electrical signal in the 2-5 cycle-per-minute (cpm) spectrum as defined by reference ranges at Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal frequency | Post meal at 3 hours
  Successful detection of gastric electrical signal in the 2-5 cycle-per-minute (cpm) spectrum as defined by reference ranges at Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal frequency | Post meal at 4 hours
  Successful detection of gastric electrical signal in the 2-5 cycle-per-minute (cpm) spectrum as defined by reference ranges at Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal amplitude | Pre-meal
  Estimation of the power of the gastric electrical signal in the above frequency spectrum (μV) at a Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal amplitude | Post meal at 1 hour
  Estimation of the power of the gastric electrical signal in the above frequency spectrum (μV) at a Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal amplitude | Post meal at 2 hours
  Estimation of the power of the gastric electrical signal in the above frequency spectrum (μV) at a Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal amplitude | Post meal at 3 hours
  Estimation of the power of the gastric electrical signal in the above frequency spectrum (μV) at a Reliability of 90% and Confidence Interval (CI) of 95%
Gastric electrical signal amplitude | Post meal at 4 hours
  Estimation of the power of the gastric electrical signal in the above frequency spectrum (μV) at a Reliability of 90% and Confidence Interval (CI) of 95%
Safety - abdominal skin effects | After removal of Gastric Alimetry array at approximately 4.2 hours post meal
  Incidence of skin irritation from the electrodes / adhesive, discomfort associated with device wear or removal
Safety - abdominal skin effects | 24 hours post study visit
  Incidence of skin irritation from the electrodes / adhesive, discomfort associated with device wear or removal
Safety - abdominal skin effects | 7 days post study visit
  Incidence of skin irritation from the electrodes / adhesive, discomfort associated with device wear or removal
Upper Gastric Symptoms - nausea, bloating, upper gut pain, heartburn, stomach burn, excessively full | Pre-meal
  Self reported assessment of symptoms on a scale of 0-10 with 10 being most severe imaginable
Upper Gastric Symptoms - nausea, bloating, upper gut pain, heartburn, stomach burn, excessively full | Post meal at 1 hour
  Self reported assessment of symptoms on a scale of 0-10 with 10 being most severe imaginable
Upper Gastric Symptoms - nausea, bloating, upper gut pain, heartburn, stomach burn, excessively full | Post meal at 2 hours
  Self reported assessment of symptoms on a scale of 0-10 with 10 being most severe imaginable
Upper Gastric Symptoms - nausea, bloating, upper gut pain, heartburn, stomach burn, excessively full | Post meal at 3 hours
  Self reported assessment of symptoms on a scale of 0-10 with 10 being most severe imaginable
Upper Gastric Symptoms - nausea, bloating, upper gut pain, heartburn, stomach burn, excessively full | Post meal at 4 hours
  Self reported assessment of symptoms on a scale of 0-10 with 10 being most severe imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Andrews, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada